CLINICAL TRIAL: NCT00369317
Title: The Treatment of Down Syndrome Children With Acute Myeloid Leukemia (AML) and Myelodysplastic Syndromes (MDS) Under the Age of 4 Years
Brief Title: Combination Chemotherapy in Treating Young Patients With Down Syndrome and Acute Myeloid Leukemia or Myelodysplastic Syndromes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAML0431; NCI-2009-00318 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000492776 (Other: Clinical Trials.gov); COG-AAML0431 (Other: Children's Oncology Group); AAML0431 (Other: CTEP); U10CA098543 (NIH)
Record Dates: First submitted 2006-08-24; First posted 2006-08-29 (Estimated); Results first posted 2015-01-13 (Estimated); Last update posted 2022-01-28 (Actual); Status verified 2021-03

CONDITIONS: Childhood Acute Basophilic Leukemia; Childhood Acute Eosinophilic Leukemia; Childhood Acute Erythroleukemia (M6); Childhood Acute Megakaryocytic Leukemia (M7); Childhood Acute Minimally Differentiated Myeloid Leukemia (M0); Childhood Acute Monoblastic Leukemia (M5a); Childhood Acute Monocytic Leukemia (M5b); Childhood Acute Myeloblastic Leukemia With Maturation (M2); Childhood Acute Myeloblastic Leukemia Without Maturation (M1); Childhood Acute Myelomonocytic Leukemia (M4); Childhood Myelodysplastic Syndromes; de Novo Myelodysplastic Syndromes; Secondary Acute Myeloid Leukemia; Secondary Myelodysplastic Syndromes; Untreated Childhood Acute Myeloid Leukemia and Other Myeloid Malignancies
MeSH Terms: conditions — Leukemia, Eosinophilic, Acute | interventions — Asparaginase; palmitoyl-L-asparaginase; Daunorubicin; Cytarabine; Thioguanine; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (combination chemotherapy) (Experimental): INDUCTION THERAPY COURSE I: Patients receive cytarabine IT on day 1 and cytarabine IV continuously over 96 hours, daunorubicin hydrochloride IV continuously, and oral thioguanine BID on days 1-4. COURSE II: Patients receive high-dose cytarabine IV over 3 hours BID on days 1, 2, 8, and 9 and asparaginase (IM) on days 2 and 9.
  COURSE III: Patients receive treatment as in course I. COURSE IV: Patients receive cytarabine IV, daunorubicin hydrochloride IV, and oral thioguanine as in course I
  INTENSIFICATION THERAPY: Patients receive cytarabine IV continuously over 168 hours on days 1-7 and etoposide IV over 1 hour on days 1-3. Treatment repeats every 28 days for 2 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: asparaginase; Drug: daunorubicin hydrochloride; Drug: cytarabine; Drug: thioguanine; Drug: etoposide; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: asparaginase — Given IM
  Other Names: ASNase; Colaspase; Crasnitin; Elspar; L-ASP
Drug: daunorubicin hydrochloride — Given IV
  Other Names: Cerubidin; Cerubidine; daunomycin hydrochloride; daunorubicin; RP-13057
Drug: cytarabine — Given IV or IT
  Other Names: ARA-C; arabinofuranosylcytosine; arabinosylcytosine; Cytosar-U; cytosine arabinoside
Drug: thioguanine — Given orally
  Other Names: 6-TG
Drug: etoposide — Given IV
  Other Names: EPEG; VP-16; VP-16-213
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase III trial is studying how well combination chemotherapy works in treating young patients with Down syndrome and acute myeloid leukemia or myelodysplastic syndromes. Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the event-free survival (EFS) and overall survival rates in pediatric patients with Down syndrome (DS) and acute myeloid leukemia AML or myelodysplastic syndromes MDS treated with induction therapy comprising cytarabine, daunorubicin hydrochloride, thioguanine, and asparaginase followed by intensification therapy comprising cytarabine and etoposide.

II. Determine if the EFS rate in these patients can be increased with an intensified course of cytarabine therapy during induction therapy, compared to the EFS rate of patients in protocol COG-A2971.

III. Determine if the number of intrathecal chemotherapy treatments can be reduced in these patients.

IV. Determine if the total cumulative anthracycline dose can be reduced in these patients.

SECONDARY OBJECTIVES:

I. Determine the type and degree of treatment-related toxicity in these patients.

II. Determine the prevalence of leukemia phenotype and globin transcription factor 1 (GATA1) mutations of DS patients < 4 years of age at diagnosis.

III. Determine the relationship of GATA1 mutations with leukemia phenotype and EFS rates of DS patients < 4 years of age at diagnosis.

IV. Determine the relationship of minimal residual disease monitored by flow cytometry and remission status during and after completion of therapy based on bone marrow morphology.

V. Examine parameters of in vitro drug sensitivity and in vivo Ara-C pharmacokinetics.

VI. Examine gene expression profiles by microarrays and the relationship to leukemia phenotype and outcome.

VII. Examine the relationship of functional polymorphisms in phase I and phase II detoxification genes and DNA repair pathways that may modify susceptibility to leukemia and outcome of therapy in DS children.

VIII. Assess the effect of karyotypic abnormalities on survival. IX. Establish a DS leukemia cell bank for future biological studies.

OUTLINE: This is a nonrandomized, multicenter study.

INDUCTION THERAPY: Patients undergo 4 courses of induction therapy. Each course is 28 days.

COURSE I: Patients receive intrathecal (IT) cytarabine on day 1* and cytarabine IV continuously over 96 hours, daunorubicin hydrochloride IV continuously over 96 hours, and oral thioguanine twice daily on days 1-4.

NOTE: *Patients with Central Nervous System (CNS) disease receive cytarabine IT twice weekly for up to 6 doses; patients with persistent CNS leukemia after 6 doses of IT cytarabine are removed from the study.

COURSE II: Patients receive high-dose cytarabine IV over 3 hours twice daily on days 1, 2, 8, and 9 and asparaginase intramuscularly (IM) on days 2 and 9.

COURSE III: Patients receive treatment as in course 1.

COURSE IV: Patients receive cytarabine IV, daunorubicin hydrochloride IV, and oral thioguanine as in course 1.

Induction therapy continues in the absence of disease progression or unacceptable toxicity. Patients with partial response, relapsed, or refractory disease after completion of course 4 are taken off study. Patients achieving complete response proceed to intensification therapy.

INTENSIFICATION THERAPY: Patients receive cytarabine IV continuously over 168 hours on days 1-7 and etoposide IV over 1 hour on days 1-3. Treatment repeats every 28 days for 2 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically for 5 years and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis DS or DS mosaicism by karyotype or chromosomal analysis
* Diagnosis of myelodysplastic syndromes (MDS) with < 30% blasts or acute myeloid leukemia (AML)

  * Newly diagnosed disease
* Patients with a history of transient myeloproliferative disorder (TMD) are eligible provided the patient is diagnosed with AML or MDS at > 90 days of age AND meets either of the following criteria:

  * At least 30% blasts in the bone marrow regardless of time since resolution of TMD
  * More than 8 weeks since resolution of TMD with ≥ 5% blasts in the bone marrow
* Immunophenotype required for study entry
* No promyelocytic leukemia
* Shortening fraction ≥ 27% by echocardiogram OR ejection fraction ≥ 50% by radionuclide angiogram
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST or ALT < 2.5 times ULN
* Creatinine adjusted according to age as follows:

  * No greater than 0.4 mg/dL (≤ 5 months)
  * No greater than 0.5 mg/dL (6 months -11 months)
  * No greater than 0.6 mg/dL (1 year-23 months)
  * No greater than 0.8 mg/dL (2 years-5 years)
  * No greater than 1.0 mg/dL (6 years-9 years)
  * No greater than 1.2 mg/dL (10 years-12 years)
  * No greater than 1.4 mg/dL (13 years and over [female])
  * No greater than 1.5 mg/dL (13 years to 15 years [male])
  * No greater than 1.7 mg/dL (16 years and over [male])
* Creatinine clearance or radioisotope glomerular filtration rate at least 70 mL/min
* No evidence of dyspnea at rest
* No exercise intolerance
* Pulse oximetry > 94%
* No prior chemotherapy, radiotherapy, or any antileukemic therapy

  * Intrathecal cytarabine therapy given at diagnosis allowed
* Prior therapy for TMD allowed

Max Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 205 (Actual)
Dates: Start 2007-03; Primary Completion 2013-12-01 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Taub, MD, Principal Investigator — Children's Oncology Group
Locations (97):
- United States (88):
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Southern California Permanente Medical Group, Downey, California
  - Miller Children's Hospital, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital Central California, Madera, California
  - Children's Hospital and Research Center at Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Childrens Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - University of California San Francisco Medical Center-Parnassus, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Lombardi Comprehensive Cancer Center at Georgetown University, Washington D.C., District of Columbia
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Memorial Healthcare System - Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic - Jacksonville, Jacksonville, Florida
  - Florida Hospital, Orlando, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - University of Hawaii, Honolulu, Hawaii
  - Saint Luke's Mountain States Tumor Institute, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Advocate Lutheran General Hospital., Park Ridge, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University, Springfield, Illinois
  - Indiana University Medical Center, Indianapolis, Indiana
  - Riley Hospital for Children, Indianapolis, Indiana
  - Saint Vincent Hospital and Health Services, Indianapolis, Indiana
  - Kosair Children's Hospital, Louisville, Kentucky
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University-Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Wayne State University-Karmanos Cancer Institute, Detroit, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Helen DeVos Children's Hospital at Spectrum Health, Grand Rapids, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Medical Center-Fairview, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - The Childrens Mercy Hospital, Kansas City, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Nevada Cancer Research Foundation CCOP, Las Vegas, Nevada
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - UMDNJ - Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Ny Cancer%, Valhalla, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Sanford Medical Center-Fargo, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Emanuel Hospital and Health Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Penn State Hershey Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Palmetto Health Richland, Columbia, South Carolina
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Vermont, Burlington, Vermont
  - Childrens Hospital-King's Daughters, Norfolk, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Princess Margaret Hospital for Children, Perth, Western Australia, Australia
- Canada (7):
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Janeway Child Health Centre, St. John's, Newfoundland and Labrador
  - Cancer Centre of Southeastern Ontario at Kingston General Hospital, Kingston, Ontario
  - Children's Hospital, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
- San Jorge Children's Hospital, Santurce, Puerto Rico

REFERENCES:
- [Derived] Taub JW, Berman JN, Hitzler JK, Sorrell AD, Lacayo NJ, Mast K, Head D, Raimondi S, Hirsch B, Ge Y, Gerbing RB, Wang YC, Alonzo TA, Campana D, Coustan-Smith E, Mathew P, Gamis AS. Improved outcomes for myeloid leukemia of Down syndrome: a report from the Children's Oncology Group AAML0431 trial. Blood. 2017 Jun 22;129(25):3304-3313. doi: 10.1182/blood-2017-01-764324. Epub 2017 Apr 7. PMID 28389462
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Combination Chemotherapy): INDUCTION THERAPY COURSE I: Patients receive cytarabine IT on day 1 and cytarabine IV continuously over 96 hours, daunorubicin hydrochloride IV continuously, and oral thioguanine BID on days 1-4. COURSE II: Patients receive high-dose cytarabine IV over 3 hours BID on days 1, 2, 8, and 9 and asparaginase (IM) on days 2 and 9.
  COURSE III: Patients receive treatment as in course I. COURSE IV: Patients receive cytarabine IV, daunorubicin hydrochloride IV, and oral thioguanine as in course I
  INTENSIFICATION THERAPY: Patients receive cytarabine IV continuously over 168 hours on days 1-7 and etoposide IV over 1 hour on days 1-3. Treatment repeats every 28 days for 2 courses in the absence of disease progression or unacceptable toxicity.
  asparaginase: Given IM
  daunorubicin hydrochloride: Given IV
  cytarabine: Given IV or IT
  thioguanine: Given orally
  etoposide: Given IV
  laboratory biomarker analysis: Correlative studies
Period: Overall Study
Arm/Group | Treatment (Combination Chemotherapy)
Started | 205
Completed | 185
Not Completed | 20
Not completed — Adverse Event | 3
Not completed — Death | 1
Not completed — Lack of Efficacy | 5
Not completed — Physician Decision | 2
Not completed — Withdrawal by Subject | 8
Not completed — Ineligible | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Combination Chemotherapy)
Number analyzed (Participants) | 205
Age, Continuous [Mean (Standard Deviation); unit: days] | 616.41 (265.73)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 205
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 106
  Male | 99
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 12
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 28
  White | 141
  More than one race | 0
  Unknown or Not Reported | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 48
  Not Hispanic or Latino | 154
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 187
  Canada | 11
  Australia | 7

OUTCOME MEASURES:

1. Primary Outcome: Event-free Survival (EFS) at 3 Years
Time Frame: Time from study entry to induction failure, relapse, or death assessed at 3 years.
Population: Ineligible patients are excluded from analyses of event free survival and overall survival.
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | Treatment (Combination Chemotherapy)
Number analyzed (Participants) | 204
percentage | 90.1 [84.8 to 93.6]

2. Primary Outcome: Overall Survival (OS) at 3 Years
Time Frame: Time from study entry to death, assessed at 3 years.
Population: Ineligible patients are excluded from analyses of overall survival and event free survival.
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | Treatment (Combination Chemotherapy)
Number analyzed (Participants) | 204
percentage | 92.7 [88.0 to 95.6]

3. Secondary Outcome: Induction Remission Rate
Description: Proportion of participants with a remission after four courses of Induction therapy.
Time Frame: End of induction therapy (day 112)
Population: Ineligible (n=1) patients are excluded. Patients who withdrew from therapy before completing 4 courses of Induction and did not die or relapse are not evaluable (n=9) for Induction remission rate.
Measure: Number; unit: Proportion of participants
Arm/Group | Treatment (Combination Chemotherapy)
Number analyzed (Participants) | 195
Proportion of participants | 0.984615

4. Secondary Outcome: Percentage of Patients Experiencing Grade 3 or 4 Toxicity Assessed by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0
Description: Proportion of participants with at least one grade 3 or higher adverse event during therapy.
Time Frame: From the beginning of induction therapy to the end of intensification therapy
Population: Ineligible patients (n=1) are excluded.
Measure: Number; unit: Proportion of participants
Arm/Group | Treatment (Combination Chemotherapy)
Number analyzed (Participants) | 204
Proportion of participants | 0.911765

5. Secondary Outcome: Prevalence of Leukemia Phenotype of DS Patients < 4 Years of Age at Diagnosis by Flow Cytometry
Description: Proportion of participants having megakaryoblastic subtype (AMkL) phenotype among patients with phenotype data available.
Time Frame: At the start of therapy
Population: Ineligible patients (n=1) are excluded. Patients without available or evaluable phenotype data are excluded (n=40). Data are not available at end of therapy or relapse.
Measure: Number; unit: Proportion of participants
Arm/Group | Treatment (Combination Chemotherapy)
Number analyzed (Participants) | 164
Proportion of participants | 0.45122

6. Secondary Outcome: Prevalence of of GATA1 Mutations of DS Patients < 4 Years of Age at Diagnosis
Description: Proportion of participants having GATA1 mutation among patients with phenotype data available.
Time Frame: At baseline and at the end of therapy (intensification) or disease relapse
Population: Ineligible patients (n=1) are excluded. Patients without available or evaluable phenotype data are excluded (n=158). Data are not available at end of therapy or relapse.
Measure: Number; unit: Proportion of participants
Arm/Group | Treatment (Combination Chemotherapy)
Number analyzed (Participants) | 46
Proportion of participants | 0.891304

7. Secondary Outcome: Proportions of Patients in Morphologic Remission With Positive MRD by Flow Cytometry
Description: Proportion of participants in complete remission by morphology and with positive MRD by flow cytometry among patients having evaluable remission and MRD assessment.
Time Frame: After Induction I therapy (day 28 from start of therapy)
Population: Ineligible patients (n=1) are excluded. Patients without available MRD at end of Induction I (n=58) or not evaluable for morphologic remission assessment (n=7) are excluded. MRD data are not available at end of Induction IV or after completion of Intensification therapy.
Measure: Number; unit: Proportion of participants
Arm/Group | Treatment (Combination Chemotherapy)
Number analyzed (Participants) | 139
Proportion of participants | 0.0935254

8. Secondary Outcome: Cytarabine Drug Sensitivity by R-Strip (MicroMath) Curve Fitting Program
Description: Mean and standard deviation of peak plasma concentration. Specimen draws were performed only with dose 1, day 1 of induction II of AraC. First sample drawn pre-infusion, then drawn 30 mins prior to the end of the infusion, and then drawn for 6 time periods post infusion up to 8 hours post infusion (and before the 2nd dose of AraC). Results are based from these multiple time points on Day 1 of Induction II only.
Time Frame: Days 1, 2, 8, and 9 of induction II
Population: Ineligible patients (n=1) are excluded. Patients without available data from peak plasma concentration (n=146) are excluded.
Measure: Mean (Standard Deviation); unit: Mean micromolar
Arm/Group | Treatment (Combination Chemotherapy)
Number analyzed (Participants) | 58
Mean micromolar | 32.69931 (18.545798)

9. Secondary Outcome: Cytarabine Drug Sensitivity by R-Strip (MicroMath) Curve Fitting Program
Description: Mean and standard deviation of area under the concentration time curve. Specimen draws were performed only with dose 1, day 1 of induction II of AraC. First sample drawn pre-infusion, then drawn 30 mins prior to the end of the infusion, and then drawn for 6 time periods post infusion up to 8 hours post infusion (and before the 2nd dose of AraC). Results are based from these multiple time points on Day 1 of Induction II only.
Time Frame: Days 1, 2, 8, and 9 of induction II
Population: Ineligible patients (n=1) are excluded. Patients without available data for area under the concentration time curve (n=146) are excluded.
Measure: Mean (Standard Deviation); unit: Mean micromolar x minutes
Arm/Group | Treatment (Combination Chemotherapy)
Number analyzed (Participants) | 58
Mean micromolar x minutes | 1337.279 (1172.20853)

10. Secondary Outcome: Cytarabine Drug Sensitivity by R-Strip (MicroMath) Curve Fitting Program
Description: Mean and standard deviation of half-life of elimination. Specimen draws were performed only with dose 1, day 1 of induction II of AraC. First sample drawn pre-infusion, then drawn 30 mins prior to the end of the infusion, and then drawn for 6 time periods post infusion up to 8 hours post infusion (and before the 2nd dose of AraC). Results are based from these multiple time points on Day 1 of Induction II only.
Time Frame: Days 1, 2, 8, and 9 of induction II
Population: Ineligible patients (n=1) are excluded. Patients without available data for half-life of elimination (n=146) are excluded.
Measure: Mean (Standard Deviation); unit: Mean minutes
Arm/Group | Treatment (Combination Chemotherapy)
Number analyzed (Participants) | 58
Mean minutes | 306.156034 (307.042662)

11. Secondary Outcome: Gene Expression Profiles by Microarrays
Description: A hierarchical clustering algorithm is used to assemble the genes into a dendrogram or tree structure with branches containing genes with similar patterns of expression. This ordered representation can be graphically displayed with colors that reflect the qualitative and quantitative relationships of the expressed genes.
Time Frame: At baseline and at the time of relapse (if available)
Population: The Microarray analysis secondary outcome is not available because the number of specimens with good quality wasn't sufficient to yield meaningful results.
Arm/Group | Treatment (Combination Chemotherapy)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: SAE field contains NCI CTCAEs submitted via expedited reporting (NCI AdEERs / CAeRs). The AE field contains grade 3 and higher CTCAEs reported on study excluding those that were reported as SAEs.
Arm/Group | Treatment (Combination Chemotherapy)
Serious Adverse Events (participants affected / at risk) | 3/204
Other Adverse Events (participants affected / at risk) | 185/204
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Combination Chemotherapy) (N=204)
Ascites (Gastrointestinal disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Immune system disorders - Other (Immune system disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1
Typhlitis (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Combination Chemotherapy) (N=204)
Abdominal pain (Gastrointestinal disorders) | 2
Acidosis (Metabolism and nutrition disorders) | 4
Activated partial thromboplastin time prolonged (Investigations) | 2
Acute kidney injury (Renal and urinary disorders) | 1
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2
Alanine aminotransferase increased (Investigations) | 23
Alkalosis (Metabolism and nutrition disorders) | 1
Anal pain (Gastrointestinal disorders) | 1
Anaphylaxis (Immune system disorders) | 5
Anemia (Blood and lymphatic system disorders) | 2
Anorectal infection (Infections and infestations) | 1
Anorexia (Metabolism and nutrition disorders) | 24
Apnea (Respiratory, thoracic and mediastinal disorders) | 1
Aspartate aminotransferase increased (Investigations) | 9
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2
Bladder infection (Infections and infestations) | 1
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 1
Blood bilirubin increased (Investigations) | 1
Cardiac arrest (Cardiac disorders) | 1
Cardiac disorders - Other (Cardiac disorders) | 4
Catheter related infection (Infections and infestations) | 22
Colitis (Gastrointestinal disorders) | 4
Conjunctivitis infective (Infections and infestations) | 1
Dehydration (Metabolism and nutrition disorders) | 4
Device related infection (Infections and infestations) | 1
Diarrhea (Gastrointestinal disorders) | 18
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Electrocardiogram QT corrected interval prolonged (Investigations) | 4
Encephalopathy (Nervous system disorders) | 1
Endocarditis infective (Infections and infestations) | 1
Enterocolitis infectious (Infections and infestations) | 13
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Esophagitis (Gastrointestinal disorders) | 1
Eye infection (Infections and infestations) | 1
Fatigue (General disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 105
Fever (General disorders) | 7
Gastritis (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1
GGT increased (Investigations) | 3
Gum infection (Infections and infestations) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 13
Hyperkalemia (Metabolism and nutrition disorders) | 8
Hypertension (Vascular disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 3
Hypocalcemia (Metabolism and nutrition disorders) | 11
Hypoglycemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 17
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 7
Hypophosphatemia (Metabolism and nutrition disorders) | 5
Hypotension (Vascular disorders) | 8
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 21
Infections and infestations - Other (Infections and infestations) | 122
Investigations - Other (Investigations) | 1
Irritability (General disorders) | 1
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 1
Lipase increased (Investigations) | 2
Lung infection (Infections and infestations) | 12
Lymphocyte count decreased (Investigations) | 2
Malabsorption (Gastrointestinal disorders) | 1
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 20
Nausea (Gastrointestinal disorders) | 1
Nervous system disorders - Other (Nervous system disorders) | 1
Neutrophil count decreased (Investigations) | 13
Oral hemorrhage (Gastrointestinal disorders) | 1
Oral pain (Gastrointestinal disorders) | 5
Otitis externa (Infections and infestations) | 1
Otitis media (Infections and infestations) | 2
Pain (General disorders) | 6
Pain of skin (Skin and subcutaneous tissue disorders) | 1
Pericardial effusion (Cardiac disorders) | 2
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1
Photophobia (Eye disorders) | 1
Platelet count decreased (Investigations) | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2
Purpura (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1
Seizure (Nervous system disorders) | 1
Sepsis (Infections and infestations) | 8
Serum amylase increased (Investigations) | 1
Sinus tachycardia (Cardiac disorders) | 2
Sinusitis (Infections and infestations) | 1
Skin infection (Infections and infestations) | 7
Small intestine infection (Infections and infestations) | 2
Soft tissue infection (Infections and infestations) | 2
Stridor (Respiratory, thoracic and mediastinal disorders) | 1
Typhlitis (Gastrointestinal disorders) | 2
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Upper respiratory infection (Infections and infestations) | 11
Urinary tract infection (Infections and infestations) | 6
Vascular access complication (Injury, poisoning and procedural complications) | 1
Vomiting (Gastrointestinal disorders) | 8
Vulval infection (Infections and infestations) | 1
Weight loss (Investigations) | 1
White blood cell decreased (Investigations) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior Sponsor approval.